CLINICAL TRIAL: NCT02308150
Title: Evaluation of Clinical Outcomes of Transcatheter Aortic Valve Replacement in the Asian Pacific Population
Brief Title: The Asian Transcatheter Aortic Valve Replacement Registry
Acronym: Asian TAVR
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2014-14
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Aortic Valve Stenosis; Aortic Diseases
Keywords: transcatheter aortic valve replacement; asian pacific; asian
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Diseases | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: transcatheter aortic valve replacement
  Other Names: TAVR

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes of transcatheter aortic valve replacement (TAVR) in the Asian Pacific population

DETAILED DESCRIPTION:
This registry changes to TP-TAVR registry(NCT03826264). Some subjects moved to TP-TAVR registry and continue to 10-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic severe aortic stenosis who are not candidates for surgical aortic valve replacement because of coexisting illnesses
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who will undergo TAVR in Asian Pacific countries
Sampling Method: Probability Sample
Enrollment: 1505 (Actual)
Dates: Start 2014-12; Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Death | 1 month
Death | 6 months
Death | 1 year
Death | 2 years
Death | 3 years
Death | 4 years
Death | 5 years

SECONDARY OUTCOMES:
Death from cardiac cause | 1 month
Death from cardiac cause | 6 months
Death from cardiac cause | 1 year
Death from cardiac cause | 2 years
Death from cardiac cause | 3 years
Death from cardiac cause | 4 years
Death from cardiac cause | 5 years
Stroke | 1 month
Stroke | 6 months
Stroke | 1 year
Stroke | 2 years
Stroke | 3 years
Stroke | 4 years
Stroke | 5 years
Myocardial infarction | 1 month
Myocardial infarction | 6 months
Myocardial infarction | 1 year
Myocardial infarction | 2 years
Myocardial infarction | 3 years
Myocardial infarction | 4 years
Myocardial infarction | 5 years
Repeat hospitalization | 1 month
Repeat hospitalization | 6 months
Repeat hospitalization | 1 year
Repeat hospitalization | 2 years
Repeat hospitalization | 3 years
Repeat hospitalization | 4 years
Repeat hospitalization | 5 years
Acute kidney injury | 1 month
Acute kidney injury | 6 months
Acute kidney injury | 1 year
Acute kidney injury | 2 years
Acute kidney injury | 3 years
Acute kidney injury | 4 years
Acute kidney injury | 5 years
Vascular complication | 1 month
Vascular complication | 6 months
Vascular complication | 1 year
Vascular complication | 2 years
Vascular complication | 3 years
Vascular complication | 4 years
Vascular complication | 5 years
Bleeding events | 1 month
Bleeding events | 6 months
Bleeding events | 1 year
Bleeding events | 2 years
Bleeding events | 3 years
Bleeding events | 4 years
Bleeding events | 5 years
Device success | 1 month
Device success | 6 months
Device success | 1 year
Device success | 2 years
Device success | 3 years
Device success | 4 years
Device success | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, Principal Investigator — Asan Medical Center; Paul Hsien Li Kao, MD, Principal Investigator — National Taiwan University; Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital, Japan; Gerald Yong, MD, Principal Investigator — Royal Perth Hospital, Australia; Kentaro Hayashida, MD, Principal Investigator — Keio University, JAPAN
Locations (12):
- Queen Elizabeth Hospital, Hong Kong, China
- Japan (5):
  - Shonan Kamakura General Hospital, Kamakura
  - Kokura Memorial Hospital, Kitakyushu
  - Keio University, Minato
  - Teikyo University School of medicine, Tokyo
  - Saiseikai Yokohama-city Eastern Hospital, Yokohama
- National University Heart Centre, Singapore, Singapore
- South Korea (4):
  - Asan Medical Center, Seoul, Songpa-gu
  - Sejong Hospital, Bucheon-si
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.

REFERENCES:
- [Derived] Yoon SH, Ahn JM, Hayashida K, Watanabe Y, Shirai S, Kao HL, Yin WH, Lee MK, Tay E, Araki M, Yamanaka F, Arai T, Lin MS, Park JB, Park DW, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Muramatsu T, Hanyu M, Kozuma K, Kim HS, Saito S, Park SJ; Asian TAVR Investigators. Clinical Outcomes Following Transcatheter Aortic Valve Replacement in Asian Population. JACC Cardiovasc Interv. 2016 May 9;9(9):926-33. doi: 10.1016/j.jcin.2016.01.047. PMID 27151607